CLINICAL TRIAL: NCT00770380
Title: Hypnosis for Smoking Relapse Prevention
Acronym: HypnoRelapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16RT-0074; 18109-557309 (Other: TRDRP)
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Smoking
Keywords: smoking
MeSH Terms: conditions — Smoking | interventions — Secondary Prevention; Hypnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hypnosis for relapse prevention (Experimental): The hypnosis intervention was conducted in two face-to-face visits with hypnosis recorded for home practice. Learning, practicing, and employing hypnotic skills in resisting the urge to smoke are core components of this intervention.
  Interventions: Other: hypnosis for relapse prevention
- Behavioral relapse prevention counseling (Active Comparator): In the behavioral relapse prevention counseling, participants were taught coping strategies for resisting the urge to smoke. This intervention focused on relapse prevention (i.e., maintenance stage of change) and was based on the theoretical concepts and treatment procedures advocated by Marlatt and Gordon and recent smoking relapse data.
  Interventions: Behavioral: behavioral relapse prevention counseling

INTERVENTIONS:
Behavioral: behavioral relapse prevention counseling — Behavioral relapse prevention counseling conducted in two one-hour sessions
  Other Names: relapse prevention
  Arms: Behavioral relapse prevention counseling
Other: hypnosis for relapse prevention — Hypnosis for relapse prevention conducted in two one-hour sessions
  Other Names: hypnotherapy
  Arms: Hypnosis for relapse prevention

SUMMARY:
A majority of smokers who quit return to smoking within three months of their quit date. This study is a randomized trial to investigate the effectiveness of hypnosis versus behavioural counseling to promote maintenance of abstinence or relapse prevention in quitting smokers. The hypothesis is that hypnosis will be at least as effective as behavioral counseling in preventing relapse to smoking in smokers who are able to quit for at least three days.

DETAILED DESCRIPTION:
We will enroll 520 current smokers in the study. All subjects will participate in an initial smoking cessation intervention involving brief counseling and nicotine replacement therapy. Participants who are able to achieve at least 3 consecutive days of abstinence will be randomized to one of two relapse prevention interventions. The participants in Study Arm 1 will receive a hypnosis intervention designed to facilitate relapse prevention. Participants in Study Arm 2 will participate in empirically-supported behavior relapse prevention counseling, utilizing the National Cancer Institute's Forever Free materials. Both interventions will be conducted in two 60-minute individual sessions scheduled one week apart in addition to counseling phone calls on their quit date and after relapse prevention treatment.

Outcomes for the two study arms will be compared by assessing biochemically-validated point-prevalence smoking status at 9 weeks(end of treatment), 26 weeks and 52 weeks. Hypnosis for relapse prevention is designed to sustain the ex-smokers commitment to remain abstinent, to provide a review of behavioral skills to resist the temptations to smoke, and to encourage attempts to quit again if relapse occurs.

ELIGIBILITY:
Inclusion Criteria:

* currently smoking at least 5/cigarettes per day during the past week
* willingness to participate and give informed consent
* aged 18 and above

Exclusion Criteria:

* contraindications to nicotine replacement
* pregnancy, lactation
* unstable psychiatric disorders
* current (last 3 months)substance use disorder
* terminal illness
* current use of smoking cessation medication

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2007-06; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Point prevalence smoking status at 9, 26 and 52 weeks | one year
  Point prevalence smoking status during past 7 days

SECONDARY OUTCOMES:
continuous quitting as measured by reported non-smoking at 9, 26 and 52 weeks continuously | one year
  Reported continuous abstinence from smoking

CONTACTS AND LOCATIONS:
Overall Officials: Timothy P Carmody, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Veterans Affairs Medical Center, 4150 Clement Street, San Francisco, California, United States